CLINICAL TRIAL: NCT04899024
Title: Optimizing PrEP Adherence in Sexual Minority Men Who Use Stimulants
Brief Title: PrEP Affect Regulation Treatment Innovation
Acronym: PARTI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: University of California, San Francisco (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adam Carrico, PhD, Professor and Chair, Florida International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20200231; R01DA051848 (NIH)
Record Dates: First submitted 2021-05-07; First posted 2021-05-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Medication Adherence; HIV Prevention; Stimulant Use
Keywords: Sexual Minority Men; HIV; PrEP Adherence; Contingency Management
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PARTI and CM (Contingency Management) (Experimental): The PARTI intervention will be delivered in five individual sessions during a 12-week contingency management protocol for PrEP adherence
  Interventions: Behavioral: PARTI; Behavioral: Contingency Management for PrEP Adherence
- Attention-Control and CM (Contingency Management) (Active Comparator): The attention-control condition will consist of five individual sessions where participants complete self-report measures and neutral writing exercises during a 12-week contingency management protocol for PrEP adherence
  Interventions: Behavioral: Attention-Control; Behavioral: Contingency Management for PrEP Adherence

INTERVENTIONS:
Behavioral: PARTI — PARTI will provide positive affect skills. Each 1-hour session delivered via Zoom consists of a didactic portion with in vivo skills practice and participants are asked to complete home practice of the skills between sessions. Many sessions include formal exercises that have been utilized in Mindfulness-Based Relapse Prevention to cultivate mindfulness and meta-cognitive awareness.
  Arms: PARTI and CM (Contingency Management)
Behavioral: Attention-Control — Attention-Control will provide a core set of coping and affect measures as well as neutral writing exercises. Each 1-hour attention-control session will be administered via Zoom.
  Arms: Attention-Control and CM (Contingency Management)
Behavioral: Contingency Management for PrEP Adherence — Participants will complete a 12-week contingency management protocol via their smartphone that consists of uploading brief videos taking PrEP medications up to four times per week. Total possible contingency management incentive for completing 48 observed PrEP doses is $360.

SUMMARY:
This multi-site randomized controlled trial enrolling sexual minority men who use stimulants and are currently taking pre-exposure prophylaxis (PrEP). This randomized controlled trial will test the efficacy of a PrEP Affect Regulation Treatment Innovation (PARTI) condition comprised of a 5-session positive affect intervention delivered during smartphone-based Contingency Management (CM) for directly observed PrEP doses (PARTI+CM) compared to an attention-control condition delivered during CM. The primary outcome is HIV acquisition risk measured using a combination of tenofovir-diphosphate levels in dried blood spots that are indicative of sub-optimal adherence to PrEP and recent condomless anal sex.

ELIGIBILITY:
Inclusion Criteria:

* Assigned male at birth
* Identifies as male
* Age 18 or older
* Reads and speaks English
* Reports condomless anal sex (CAS) with men in the past 6 months
* self-reported HIV negative
* Active prescription for daily oral PrEP for at least 2 months and reports any non-adherence in the past month OR initiated daily oral PrEP in the past 2 months, regardless of self-reported adherence
* Has an iPhone or Android smartphone
* Screens positive for a moderate or severe stimulant use disorder with an abbreviated version of the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST; total score of 4 or more) OR reports using stimulants at least weekly in the past 3 months.
* Lives in California or Florida with no plans to move out of state in the next 6 months

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Unwilling to upload upload 3 video recordings of directly observed PrEP doses using a smartphone application
* Identifies as transfeminine (e.g., transgender woman)
* Unable or Unwilling to provide dried blood spot (DBS) specimen at baseline
* Switched from daily oral PrEP with disoproxil fumarate (TDF) to daily oral PrEP with tenofovir alafenamide (TAF) in the past 5 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned male at birth and identifies as male.
Enrollment: 239 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2026-02-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Engaging HIV Acquisition Risk | Up to 12 months
  Percentage of participants engaging in HIV acquisition risk (i.e., defined as tenofovir - diphosphate levels < 700 fmol per punch from dried blood spots and any self-reported recent condomless anal sex)

SECONDARY OUTCOMES:
PrEP Persistence | Up to 12 months
  Percentage of participants who continue taking PrEP medication
Retention in PrEP Care | Up to 12 months
  Percentage of participants who report attending a medical visit with the PrEP provider in the past three months
Self-Reported Stimulant Use Severity | Up to 12 months
  The Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) provides validated composite scores indexing the severity of cocaine and amphetamine use (Mild = 0-3; Moderate = 4-26; Severe = 27 or greater).
Positive Affect | Up to 12 months
  Mean positive affect score as measured by the modified Differential Emotions Scale (Range 0-104) with higher scores being indicative of higher positive affect.

CONTACTS AND LOCATIONS:
Overall Officials: Adam W Carrico, PhD, Principal Investigator — Florida International University
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - University of Miami Miller School of Medicine, Miami, Florida

IPD SHARING:
Plan to Share IPD: No